CLINICAL TRIAL: NCT05747339
Title: The Efficacy and Safety of Tumor Treatment Vaccine in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study on the Efficacy and Mechanism of Tumor Treatment Vaccine (TTV) for Recurrent and Refractory Advanced Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY23009
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumors, Adult
Keywords: Tumor immunotherapy; Tumor vaccine; Advanced solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor treatment vaccine for patients with advanced solid tumors (Experimental): Tumor treatment vaccine(TTV) would be given deep subcutaneously in the arm or near the tumor.The check indexes are image examination (CT, MRI or PET scan) and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: tumor treatment vaccine injection

INTERVENTIONS:
Biological: tumor treatment vaccine injection — Patients will receive tumor treatment vaccine(TTV), which would be given deep subcutaneously in the arm or near the tumor.The initial dose is 1ml / week, if the reaction isn't obvious, the dose can be appropriately increased to 2.5-4.0ml / week.The interval between injections can be shortened or extended depending on the patient's condition and response.The duration of treatment should be extended as long as possible, at least 6-12 months.

SUMMARY:
This is a study of the clinical efficacy and mechanism study of tumor treatment vaccine (TTV, also known as Neo-BCV) in patients with recurrent and refractory advanced solid tumors.

DETAILED DESCRIPTION:
The study aims to explore the safety and effectiveness of Neo-BCV in the treatment of advanced solid tumors.The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years;
2. ASubjects must have histologically- or cytologically-confirmed diagnosis of advanced solid tumor(s) and have progressed on or is not eligible for available standard therapy;
3. Subjects have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
4. ECOG score of 0-2, lifespan > 12 weeks;
5. Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
6. Voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. The patient is diagnosed with central nervous system leukemia(symptoms, signs, imaging, cerebrospinal fluid);
2. White blood cell count ≥ 50×10^9/ L or patients with rapid disease progression can't be guaranteed to complete a full treatment cycle;
3. Patients with fungal, bacterial, viral or other uncontrollable infections or requiring four-level isolation treatment.
4. HIV, HBV and HCV positive;
5. Patients with diseases of the central nervous system or autoimmune central nervous system lesions, Including stroke, epilepsy, dementia;
6. Patients have myocardial infection, cardiac angiography or stents, active angina or other obvious clinical symptoms, or have cardiopathic asthma or cardiovascular lymphocytic infiltrates，within 12 months;
7. Patients are on anticoagulation or have severe coagulopathy (APTT>70);
8. Patients in any condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 2weeks prior to investigational drug administration;
9. Patients were infected with covid-19 within 2weeks prior to investigational drug administration;
10. Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
11. Subjects in other conditions that are considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief degree of tumors | The last injection
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST1.1）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
  The duration from the beginning of treatment to cancer recurrence or progression
Overall survival（OS） | 3 years
  The duration from the beginning of treatment to patient death